CLINICAL TRIAL: NCT05154240
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Oral Single and Multiple Ascending Doses, Parallel Group Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of INS018_055 in Healthy Subjects
Brief Title: A Phase 1, Evaluate the Safety, Tolerability, and Pharmacokinetics of INS018_055 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: INS018-055-001
Record Dates: First submitted 2021-11-17; First posted 2021-12-13 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, randomized, 2-part (Part A and B), first-in-human, double-blind, placebo controlled single and multiple ascending dose study designed to assess the safety, tolerability, and PK of INS018_055 when administered as oral doses to healthy subjects. Additionally, this study will investigate the impact of food on the PK of INS018_055.
  Part A (Single Ascending Dose [SAD]):
  Food Effect Assessment (Cohort 4 in Part A only):
  Part B (Multiple Ascending Dose [MAD]):
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INS018_055 (Active Comparator): oral doses of INS018_055_single dose; oral doses of INS018_055_multiple ascending dose over 10days.
  Interventions: Drug: INS018_055
- Placebo (Placebo Comparator): No active ingredient. Frequency similar to the 2 arms above.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INS018_055 — INS018_055 is a small molecule compound. INS018_055 has good solubility in water and was chemically and physically stable at different temperatures.
  Arms: INS018_055
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The sponsor is planning to conduct a Phase 1, randomized, double-blind, placebo-controlled, oral single and multiple ascending-doses, parallel group study to evaluate the safety, tolerability and PK of INS018_055 in healthy subjects. The study will be conducted in 1 clinical site in the New Zealand, consisting of 2 parts: Part A (single ascending dose [SAD]) and Part B (multiple ascending dose [MAD]).

DETAILED DESCRIPTION:
This is a Phase 1, randomized, 2-part (Part A and B), double-blind, placebo controlled single and multiple ascending doses study designed to assess the safety, tolerability, and PK of INS018_055 when administered as oral doses to healthy subjects. Additionally, this study will investigate the impact of food on the PK of INS018_055.

Part A (Single Ascending Dose [SAD]):

Eight healthy subjects will be assigned to each of up to 5 sequential dose cohorts and will be randomly assigned within each dose cohort to receive INS018_055 or a matched placebo in a ratio of 3:1 (6 active, 2 placebo) on Day 1 for a total of up to approximately 40 subjects. Subjects in Part A will be admitted to the study site on Day -1 and dosed on Day 1 after fasting (nothing to eat or drink, except water) for at least 10 hours. Water is not allowed 1 hour prior to and 1 hour after dosing. Water can be consumed ad libitum at other times. Subjects will remain fasted on Day 1 for 4 hours after dosing. Subjects will be discharged from the study site on Day 4, after the scheduled procedures and review of the Day 4 safety data by the investigator (or designee). Subjects will come back for an end of study (EOS) visit on Day 8 (± 1 day).

A sentinel cohort of 2 subjects will be used to mitigate the risk of unexpected adverse events (AEs) not predicted by preclinical pharmacology and toxicology studies for each dosing cohort, starting with Cohort 1 (the initial dose cohort). The sentinel subjects will be dosed in a blinded fashion (1 active, 1 placebo) and monitored for at least 1 day before the remaining 6 subjects in that cohort are dosed. Initiation of dosing of the remaining 6 subjects will depend on an initial safety review by the investigator indicating that administration of the study treatment was safe and well tolerated in the sentinel subjects.

Dose escalation will occur only after the real time PK, safety, and tolerability data (including reported AEs, physical examinations, vital signs, electrocardiograms (ECGs), and clinical laboratory results up to 48 hours after dosing) of the preceding dose cohort for at least 6 subjects are assessed and the study treatment is deemed safe and well tolerated by the safety review committee (SRC). As new safety and/or PK data become available, the anticipated dose escalation scheme may change following a review of the data by the SRC. Preliminary PK data from subjects in this study will help guide dose escalation to higher doses. Dose escalation in Cohorts 4 and 5 will only occur after the PK data from at least the first 2 cohorts have been assessed and deemed sufficient to model exposures for Cohorts 4 and 5.

Food Effect Assessment (Cohort 4 in Part A only): Subjects in Cohort 4 of Part A will participate in a food effect arm. The actual dose level for food effect cohort is subject to change and will be confirmed by the SRC after review of data from at least the first 2 cohorts of the SAD. Following the standard SAD dosing on Day 1 and at least 3 days of follow up/washout (or 5 times the estimated half-life of INS018_055 based on the observed data, whichever is longer) (Period 1), enrolled subjects will enter Period 2 and be re administered the same dose of INS018_055 or matching placebo (the same treatment that they received on Day 1 of Period 1) after completing a standard high-fat meal. Subjects will fast (nothing to eat and drink, except water) for at least 10 hours overnight and receive a standard high-fat breakfast 30 minutes prior to dosing. The high-fat breakfast will be consumed within approximately 30 minutes. Subjects will remain at the study site on Day 4 of Period 2 until the scheduled procedures and review of the Day 4 safety data by the investigator (or designee) are completed. The washout period of at least 3 days (or 5 times the estimated half life of INS018_055 based on the observed data, whichever is longer) may be extended based on available PK data from previous cohorts. The Day -1 procedures will not be repeated for Period 2.

Physical examinations, vital sign measurements, 12-lead ECGs, and clinical laboratory evaluations will be performed at selected time points throughout the study. Subjects will also be closely monitored for AEs throughout the study. Blood samples for PK will be collected up to 72 hours after study treatment administration on Day 1 for all cohorts. For biomarkers (CD4+ and CD8+ T-cells), blood samples will be collected at check-in (Day -1), Day 2, and Day 4 after administration of INS018_055. Fecal occult blood tests will be done with all stools passed at screening, check-in (Day -1), and during the 72 hour observation period. Subjects will be discharged on Day 4.

Part B (Multiple Ascending Dose [MAD]):

Eight healthy subjects will be assigned to each of up to 5 sequential once daily (QD) or twice daily (BID) dose cohorts and will be randomly assigned within each dose cohort to receive INS018_055 or a matched placebo for 10 days in a ratio of 3:1 (6 active, 2 placebo), for a total of up to approximately 40 subjects.

Subjects in Part B will begin dosing, after safety and tolerability data (including reported AEs, physical examination, clinical laboratory results, 12-lead ECGs, and vital signs) from at least the first 3 cohorts (Cohorts 1 to 3) in Part A are assessed and the study treatment is deemed safe and well tolerated by the SRC. Additionally, sufficient PK data from at least the first 3 cohorts of Part A must be obtained to model exposures in Part B. The dosing schedule, either QD or BID, will be decided by the SRC after review of the PK, safety, and tolerability data from the first 3 cohorts of Part A.

The initial MAD cohorts will begin dosing with the remaining SAD cohorts. The top dose explored in Part B will not exceed the maximum dose explored in Part A. Subsequent dose escalations in Part B will not occur until the safety (including AEs, physical examination, clinical laboratory results, vital signs, and 12-lead ECGs) and tolerability data up to and including Day 14 of the preceding MAD dose cohort for at least 6 subjects are assessed and the study treatment is deemed safe by the SRC.

As new safety or PK data become available, the dose escalation scheme may change. Subjects may not receive a subsequent higher dose and may instead be administered a lower dose or may repeat the same daily dose with a different administration schema, eg, BID instead of QD dosing, to achieve lower maximum observed plasma concentration (Cmax) values, particularly if the safety findings are believed to be linked to the Cmax values.

The highest dose in the MAD (either QD or BID) will be dosed in a staggered way if accrued PK data from previous cohorts predict potential exposures above the no observed adverse effect level, with 2 subjects starting dosing at least 7 days before the remaining 6 subjects; initiation of dosing of the remaining 6 subjects will depend on an initial safety review by the investigator indicating that administration of the study treatment was safe and well tolerated in the sentinel subjects.

Each subject in Part B will be admitted to the study site on Day -1 and will begin daily dosing on Day 1. Study treatment is to be administered daily at approximately the same time in the morning. For BID dosing, the second dose of study treatment will be administered approximately 12 hours after the morning dose of study treatment.

Prior to the morning dosing on Days 1 and 10 for Cohorts 6 to 10, subjects will fast (nothing to eat and drink, except water) for at least 10 hours overnight and remain fasted for 4 hours after study treatment administration. Water is not allowed 1 hour prior to and 1 hour after dosing. Water can be consumed ad libitum at other times. Water is not restricted for the evening doses when study treatment is being dosed BID. On Days 1 and 10, lunch will be provided approximately 4 hours after the morning dose, dinner will be provided approximately 10 hours after the morning dose, and a snack will be provided approximately 13 hours after the morning dose.

On Days 2 to 9 for Cohorts 6 to 10, breakfast will be provided approximately 60 minutes after study treatment administration. Standardized meals will be provided to the subjects throughout the study. Lunch will be provided approximately 4 hours after the morning dose, dinner will be provided approximately 10 hours after the morning dose, and a snack will be provided approximately 13 hours after the morning dose.

Physical examinations, vital sign measurements, 12-lead ECGs, and clinical laboratory evaluations (including liver function test results) will be performed at selected time points throughout the dosing interval. Subjects will be closely monitored for AEs throughout the study. Blood samples for PK analyses will be collected up to 72 hours after study treatment administration on Day 10. Urine samples for PK analysis will be collected before dosing (Day 1 as a single void collected within 0 to 24 hours) and over the following intervals after dosing: 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hours on Day 1 and 0 to 4, 4 to 8, 8 to 12, 12 to 24, and 24 to 48 hours on Day 10 for both QD and BID cohorts. For biomarkers (CD4+ and CD8+ T-cells), blood samples will be collected at selected time points for QD and BID dosing cohorts. Fecal occult blood tests will be done with all stool samples at screening, check-in (Day 1), and throughout Part B on site observation periods, ie, up to Day 14.

Subjects will be discharged from the study site on Day 14, after the scheduled procedures and review of the safety data by the investigator (or designee). Subjects will return to the study site on Day 28 (± 3 days) for an EOS visit.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or female 18 to 55 years of age, inclusive.
2. The subject has a body mass index 18 to 32 kg/m2, inclusive, and a total body weight ≥50 kg, inclusive, at screening.
3. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
4. Female subjects of childbearing potential must be non-pregnant and non-lactating and must use one of the methods of contraception listed below for the duration of the treatment until at least 28 days after the last dose of the study drug, or be surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or postmenopausal (defined as amenorrhea 12 consecutive months and documented plasma follicle stimulating hormone level >40 IU/mL). Female subjects must have a negative pregnancy test at screening and before the first dose of study drug.

   Highly effective methods of contraception are those that result in a failure rate of less than 1% per year when used consistently. Examples are provided below:
   1. Implant contraceptive (eg, Jadelle®)
   2. Intrauterine device containing either copper or levonorgestrel (eg, Mirena®)
   3. Male sterilization with absence of sperm in the post-vasectomy ejaculate

      OR an effective method that result in a failure rate of less than 5% to 10% per year. Examples are provided below:
   4. Injectable contraceptive (eg, Depo Provera)
   5. Oral contraceptive pill (combined hormonal contraceptive pill or progestogen-only 'mini-pill')
   6. Vaginal contraceptive ring (eg, NuvaRing®)

   Female subjects must also agree not to donate eggs, from dosing until at least 28 days after the last dose of study drug.

   A male subject and his female partner who is of childbearing potential must agree to use one of the methods of contraception listed above for the duration of the treatment until at least 28 days after the last dose of the study drug. A male subject must also agree not to donate sperm, for the duration of the treatment until at least 28 days after the last dose of the study drug.
5. The subject agrees to comply with all protocol requirements.
6. The subject is able to provide written informed consent.

Exclusion Criteria:

1. The subject has current evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. The subject has any condition possibly affecting drug absorption (eg, gastrectomy).
3. The subject has a history of cancer with the exception of adequately treated basal cell or squamous cell carcinoma of the skin.
4. The subject has supine blood pressure (BP) >140 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >140 mm Hg (systolic) or >90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility at screening.
5. The subject has 12-lead ECG demonstrating corrected QT interval by Fridericia (QTcF) >450 msec, or a QRS interval >120 msec at screening. If QTcF exceeds 450 msec, or QRS interval exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF (or QRS interval) values should be used to determine the subject's eligibility.
6. The subject has ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

   1. Serum creatinine level above the upper limit of normal (ULN) or an estimated glomerular filtration rate value <80 mL/min/1.73 m2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula and the absence of protein in urine, at screening.
   2. Aspartate aminotransferase or alanine aminotransferase values more than >1.5 × ULN.
   3. Fasting glucose >110 mg/dL (6.1 mmol/L).
   4. Total bilirubin >1.5 × ULN.
   5. Hematological values outside the normal reference range for local laboratory results.
   6. Positive fecal occult blood test at screening or at check-in (Day -1).
7. The subject has any medical history of disease that has the potential to cause a rise in total bilirubin over the ULN. Subjects with borderline clinical laboratory values outside the reference range may be included in the study if the investigator deems that the values are not clinically significant.

   Note: Subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is <ULN.
8. The subject has a history of any lymphoproliferative disorder (such as Epstein Barr Virus related lymphoproliferative disorder, as reported in some subjects on immunosuppressive drugs), history of lymphoma, leukemia, myeloproliferative disorders, multiple myeloma, or signs and symptoms suggestive of current lymphatic disease.
9. The subject has a history of relevant drug and/or food allergies (ie, allergy to any study drug or excipients, or any significant food allergy that could preclude a standard diet in the clinical unit).
10. The subject has a clinically significant infection currently or within 6 months of first dose of study drug (eg, those requiring hospitalization or parenteral antimicrobial therapy or opportunistic infections within the last 6 months), or a history of chronic or recurrent infectious disease.
11. The subject has other severe acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
12. The subject has or has had symptomatic herpes zoster or herpes simplex within 12 weeks, more than one episode of local herpes zoster, or a history (single episode) of disseminated zoster.
13. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
14. The subject is a female who is pregnant or lactating.
15. The subject is a fertile male who is unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
16. The subject is unwilling or unable to comply with the lifestyle restrictions described in this protocol.
17. The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
18. The subject has a positive test result for drugs of abuse, or cotinine (indicating active current smoking) at screening or before the first dose of study drug.
19. The subject has used any prescription or over the counter medications (except paracetamol [up to 2 g per day]), including herbal supplements, within 14 days before the first dose of study drug. Nutritional supplements are allowed if unlikely to interfere with the study results and agreed by medical monitor and investigator.
20. The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or alcohol-, caffeine-, or xanthine containing products within 48 hours before the first dose of study drug.
21. The subject will have vaccination with live virus, attenuated live virus, or any live viral components within 2 weeks prior to the first dose of study drug or is to receive these vaccines at any time during treatment or within 8 weeks following completion of study treatment.
22. The subject has a positive test result for severe acute respiratory syndrome-related coronavirus 2 (SARS-CoV-2). The subject has received the Coronavirus disease 2019 (COVID-19) vaccine within 2 weeks prior to the first dose of study drug or plans to receive a COVID-19 vaccine within 12 weeks after study drug dosing or has positive test for SARS CoV 2 during screening or presence of COVID 19 symptoms within 4 weeks prior to Day -1.
23. The subject has undergone significant trauma or major surgery within 4 weeks of screening.
24. The subject has bleeding risk: genetic predisposition to bleeding, a hemorrhagic event in the 12 months before the start of screening, or abnormal laboratory coagulation parameters.
25. The subject has a first-degree relative with a hereditary immunodeficiency.
26. The subject has investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are sponsor employees including their family members are directly involved in the conduct of the study.
27. The subject has a history of alcohol abuse or drug addiction within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits) or use of alcohol 48 hours before the first dose of study drug.
28. The subject is involved in strenuous activity or contact sports within 24 hours before dosing and during the study.
29. The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
30. The subject has received study drug in another investigational study within 30 days of dosing.
31. The subject received cytochrome P450 (CYP)/ multidrug and toxin extrusion (MATE) classes of medications within 4 weeks of first dose of INS018_055 or was likely to receive CYP/MATE classes of medications during the study.
32. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events based on subjective and objective examination | 12 months
  Subjective examination refers to the participant response to standard question to elicit any medically related changes in their well-being.
  Descriptive examination refers to laboratory values as reviewed by the investigator, physical examination findings and ECG Changes, or other documents that are relevant to participant safety.
  AEs will be classified as:
  Mild: These events require minimal or no treatment and do not interfere with the subject's daily activities. Moderate: These events result in a low level of inconvenience or require minor therapeutic measures. Moderate events may cause some interference with normal functioning. Severe: These events interrupt a subject's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually incapacitating.

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
AUC from time 0 extrapolated to infinity (AUC0-inf) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
AUC from time 0 to the time of the dosing interval (To; AUC0-To) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Accumulation ratio (AR), calculated as AUC0-To (Day 10)/AUC0-To (Day 1) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
AR calculated as Cmax (Day 10)/Cmax (Day 1) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Time to reach Cmax (Tmax) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Pre-dose concentrations on Days 1 through 10 (C trough) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Average concentration on Day 1 and Day 10 (Cav) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Terminal elimination rate constant (Kel) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Terminal elimination half-life (t1/2) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Apparent total body clearance (CL/F) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Peak to trough ratio calculated as Cmax/Ctrough | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Apparent volume of distribution (Vd/F) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Metabolite-to parent ratio based on AUC calculated as AUCmetabolite/AUCparent | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Metabolite-to parent ratio based on Cmax calculated as Cmax, metabolite/Cmax, parent | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Renal clearance (CLr) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.
Total amount of drug excreted unchanged in urine from 0 to 24 hours after dosing (XU0-24) | 12 months
  * To determine the PK of INS018_055 following single and multiple oral escalating doses in healthy subjects.
  * To assess the effect of food on the PK of INS018_055 following an oral dose.

OTHER OUTCOMES:
Characterisation of CD4+ and CD8+ subpopulation of T cells after single dose and of the same after multiple oral escalating doses of INS018_055 | 12 months
  To determine the effect of single doses of INS018_055 on the circulating CD4+ and CD8+ subpopulation of T cells and the effect of multiple oral escalating doses of INS018_055 on circulating CD4+ and CD8+ subpopulation of T cells as these could be used as biomarkers for the selection of the therapeutic dose range.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Wynne, MBChB, Principal Investigator — New Zealand Clinical Research
Locations (1):
- NZCR Ltd, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No